CLINICAL TRIAL: NCT07027852
Title: My Lung Health Coach-A Virtual COPD Self-management Support Program Integrated Into the Electronic Patient Record
Acronym: MLHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Andrew Kouri, Doctor Andrew Kouri, Women's College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2025-01-13; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Copd
Keywords: COPD; Telehealth; Telemonitoring; Respiratory
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Behavioral (Experimental): Study Description: My Lung Health Coach (MLHC) is a virtual COPD education and self-management support program delivered by a Certified Respiratory Educator (CRE) over 12 weeks. The investigators have also developed a companion app to MLHC integrated into the electronic patient record that patients can access through their EPIC MyHealth app. This study will evaluate the feasibility and effectiveness of MLHC and the companion app.
  Interventions: Behavioral: My Lung Health Coach

INTERVENTIONS:
Behavioral: My Lung Health Coach — Virtual education and self-management program with companion application

SUMMARY:
Study Description: My Lung Health Coach (MLHC) is a virtual COPD education and self-management support program delivered through one-on-one sessions with a Certified Respiratory Educator (CRE) over 12 weeks. It includes six sessions that cover essential COPD topics such as: Basic COPD knowledge, Smoking cessation, Medications (inhalers, oxygen), Physical activity, Mental health and wellness, Vaccinations, Symptom self-management, Nutrition, Travel, and Long-term planning (including end-of-life care). The investigators have also developed a companion app to MLHC integrated into the electronic patient record that patients can access through their EPIC MyHealth app on the participants phones, tablets, or desktops. This study will evaluate the feasibility and effectiveness of MLHC and the companion app.

DETAILED DESCRIPTION:
My Lung Health Coach (MLHC) is a freely available evidence-based and person-centered COPD self-management program that connects people virtually with experienced certified respiratory educators (CREs) to provide structured COPD education and self-management support. MLHC was jointly developed by the Lung Health Foundation (a charitable organization focused on lung health advocacy) and academic Respirologist Dr. Andrew Kouri, with input from community members living with COPD. MLHC links community members living with COPD with certified respiratory health educators, using a person-centred approach to provide COPD education and self-management support. It is delivered virtually through one-on-one meetings offered over multiple sessions over 12 weeks. The topics covered in the program include: general COPD knowledge, smoking cessation, COPD medications (inhalers, oxygen), physical activity counselling, mental health and wellness, vaccinations, symptom self-management skills (breathing, energy management, symptom monitoring), nutrition, travel, and long-term planning (including end-of-life care).

To improve the patient experience using MLHC, the investigators have integrated the MLHC program into the Epic Care Companion app at Women's College Hospital, an interactive patient-facing app designed as an extension of the Epic electronic health record system. Using Care Companion, patients will be able to track their progress through MLHC, accomplish session-specific educational and self-management tasks, and share their progress with their Women's College healthcare teams.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have capacity to provide informed consent;
2. Must sign and date the informed consent form;
3. Stated willingness to comply with all study procedures;
4. Be diagnosed with COPD as per a WCH Respirologist
5. Be 40 years or older
6. Be a current or ex-smoker
7. Preferred but not required: have a history of at least 1 COPD exacerbation (requiring prednisone or antibiotic use, or an urgent healthcare visit of any kind) in the previous 12 months

Exclusion Criteria:

1. Experienced a COPD exacerbation in the 4 previous weeks to study enrollment
2. Co-diagnosis of asthma by a WCH Respirologist
3. Significant co-morbidities that could interfere with program participation or terminal illness
4. Unwilling to download and use the Epic Care Companion app and has a unsuitable mobile device to do this
5. Pregnancy

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility (system use): Number of patients who started program over total offered, over one year. | 1 year
  Number of patients who started program over total offered for one year.
Feasibility (system use): Number of patients who completed program over total started, over one year. | 1 year
  Number of patients who completed program over total started for one year.
Feasibility (system use): Number of providers who referred patients to the program over total Number of providers, over approximately one year. | 1 year
  Number of providers who referred patients to the program over total Number of providers, over approximately one year.
Effectiveness (clinical outcomes): Number of COPD-related outpatient visits | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Number of COPD-related outpatient visits
Effectiveness (clinical outcomes): Hospital admissions | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Hospital admissions
Effectiveness (clinical outcomes): ED visits | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  ED visits
Effectiveness (clinical outcomes): ICU admissions (at baseline will be over the previous 12 months) | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  ICU admissions (at baseline will be over the previous 12 months)
Effectiveness (clinical outcomes): COPD severity as measured by the COPD assessment test (CAT) | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  COPD severity as measured by the COPD assessment test (CAT)
Effectiveness (clinical outcomes): Medication | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Medication
Effectiveness (clinical outcomes): Referrals: pulmonary rehab | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Referrals: pulmonary rehab
Effectiveness (clinical outcomes): Referrals: smoking cessation counseling | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Referrals: smoking cessation counseling
Effectiveness (clinical outcomes): Referrals: specialist care | outcomes will be collected prior to program commencement, at program completion (3 month), and at 6-month follow-up.
  Referrals: specialist care

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kouri, MD, Principal Investigator — Womens College Hospital
Locations (1):
- Womens College Hospital, Toronto, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT07027852/Prot_000.pdf